CLINICAL TRIAL: NCT00996281
Title: A Phase 3, Open-Label, Randomized, Long-Term Comparison of the Safety and Tolerability of the TAK-491 Plus Chlorthalidone Fixed-Dose Combination vs. Olmesartan Medoxomil-Hydrochlorothiazide Fixed-Dose Combination in Subjects With Essential Hypertension
Brief Title: Safety and Tolerability of Azilsartan Medoxomil Plus Chlorthalidone Compared to Olmesartan Medoxomil Plus Hydrochlorothiazide in Participants With Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAK-491CLD_308; 2008-008260-28 (Registry Identifier: EudraCT); U1111-1111-7891 (Other: WHO)
Record Dates: First submitted 2009-10-12; First posted 2009-10-16 (Estimated); Results first posted 2012-11-12 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-10

CONDITIONS: Essential Hypertension
Keywords: Hypertensive; Blood Pressure, High; Cardiovascular disease; Vascular Disease; Drug Therapy
MeSH Terms: conditions — Essential Hypertension; Hypertension; Cardiovascular Diseases; Vascular Diseases | interventions — azilsartan medoxomil; Chlorthalidone; Olmesartan Medoxomil; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Azilsartan Medoxomil and Chlorthalidone (Experimental): Azilsartan medoxomil 40 mg and chlorthalidone 12.5 mg combination tablet, orally, once daily for up to 52 weeks.
  For participants who did not achieve target blood pressure by Week 4, titration to a maximum dose of azilsartan medoxomil 80 mg and chlorthalidone 25 mg.
  Interventions: Drug: Azilsartan medoxomil and chlorthalidone
- Olmesartan Medoxomil and Hydrochlorothiazide QD (Active Comparator): Participants in the United States:
  Olmesartan medoxomil 20 mg and hydrochlorothiazide 12.5 mg combination tablet, orally, once daily for up to 52 weeks. For participants who did not achieve target blood pressure by Week 4, titration to a maximum dose of Olmesartan medoxomil 40 mg and hydrochlorothiazide 25 mg.
  Participants in Europe:
  Olmesartan medoxomil 20 mg and hydrochlorothiazide 12.5 mg combination tablet, orally, once daily for up to 52 weeks. For participants who did not achieve target blood pressure by Week 4, titration to a maximum dose of Olmesartan medoxomil 20 mg and hydrochlorothiazide 25 mg.
  Interventions: Drug: Olmesartan medoxomil and hydrochlorothiazide

INTERVENTIONS:
Drug: Azilsartan medoxomil and chlorthalidone — Combination tablet.
  Other Names: TAK-491CLD
  Arms: Azilsartan Medoxomil and Chlorthalidone
Drug: Olmesartan medoxomil and hydrochlorothiazide — Combination tablet.
  Other Names: Benicar HCT®; Olmetec Plus®
  Arms: Olmesartan Medoxomil and Hydrochlorothiazide QD

SUMMARY:
The purpose of this study is to compare the safety and tolerability of azilsartan medoxomil plus chlorthalidone, once daily (QD), versus olmesartan medoxomil-hydrochlorothiazide in adults with essential hypertension.

DETAILED DESCRIPTION:
High Blood Pressure (Hypertension) is the most common cause of preventable death in developed nations. Uncontrolled hypertension greatly increases the risk of heart disease, brain disease, and kidney failure. As the population ages, the incidence of hypertension will continue to increase if effective preventive measures are not implemented. Despite the availability of antihypertensive agents, hypertension is not adequately controlled; only about one in three patients successfully keep blood pressure normal.

Treatment for high blood pressure includes thiazides or thiazide-like diuretics, either alone or as part of combination treatment. Chlorthalidone is a commercially available, orally administered thiazide-type diuretic agent.

TAK-491 (azilsartan) is an angiotensin II receptor blocker being evaluated by Takeda to treat patients with high blood pressure (essential hypertension).

This study will compare the safety and tolerability of azilsartan medoxomil plus chlorthalidone (TAK-491CLD) fixed-dose combination to olmesartan medoxomil-hydrochlorothiazide fixed-dose combination.

Initially patients will undergo a Screening Visit to confirm that they are eligible to participate in the study. All participants will receive the study drug for up to 52 weeks. The dose of the study drug may be gradually increased throughout the study so that a target blood pressure value can be reached for each participant.

Throughout the treatment period of the study, participants will be required to visit the research site for 11 visits. At these study visits participants will be required to undergo certain study procedures including physical examinations, vital sign measurements (blood pressure, heart rate, weight and height), electrocardiograms (monitoring of the heart), and blood and urine samples taken for clinical laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* Is treated with antihypertensive therapy and has a post-washout mean sitting clinic systolic blood pressure greater than or equal to 160 and less than or equal to 190 mm Hg on Day, or has not received antihypertensive treatment within 14 days prior to Screening and has a mean sitting clinic systolic blood pressure greater than or equal to 160 and less than or equal to 190 mm Hg at the Screening Visit and on Day 1.
* Females of childbearing potential who are sexually active agree to routinely use adequate contraception, and can neither be pregnant nor lactating from before study participation to Screening to 30 days after the last study drug dose.
* Has clinical laboratory test results within the reference range for the testing laboratory or the investigator does not consider the results to be clinically significant.
* Is willing to discontinue current antihypertensive medications up to 3 weeks before enrollment.

Exclusion Criteria:

* Has a mean clinic diastolic blood pressure (sitting, trough) greater than 119 mm Hg on Day 1.
* Has secondary hypertension of any etiology (eg, renovascular disease, pheochromocytoma, Cushing's syndrome).
* Has a recent history (within the last 6 months) of myocardial infarction, heart failure, unstable angina, coronary artery bypass graft, percutaneous coronary intervention, hypertensive encephalopathy, cerebrovascular accident or transient ischemic attack.
* Has clinically significant cardiac conduction defects (ie, third-degree atrioventricular block, sick sinus syndrome).
* Has hemodynamically significant left ventricular outflow obstruction due to aortic valvular disease.
* Has severe renal dysfunction or disease.
* Has known or suspected unilateral or bilateral renal artery stenosis.
* Has a history of cancer that has not been in remission for at least 5 years prior to the first dose of study drug.
* Has poorly-controlled type 1 or 2 diabetes mellitus at Screening.
* Has hypokalemia or hyperkalemia at Screening.
* Has an alanine aminotransferase or aspartate aminotransferase level of greater than 2.5 times the upper limit of normal, active liver disease, or jaundice at Screening.
* Has any other known serious disease or condition that would compromise safety, might affect life expectancy, or make it difficult to successfully manage and follow according to the protocol.
* Has known hypersensitivity to angiotensin II receptor blockers or thiazide-type diuretics or other sulfonamide-derived compounds.
* Has been randomized/enrolled in a previous azilsartan or azilsartan medoxomil plus chlorthalidone study.
* Currently is participating in another investigational study or has received any investigational compound within 30 days prior to Screening.
* Has a history of drug abuse or a history of alcohol abuse within the past 2 years.
* Is taking or expected to take any excluded medication, including:

  * Antihypertensive medications must be discontinued completely by Day -14, except antihypertensive medications used in the open-label treatment period in accordance with the titration-to-target blood pressure titration.
  * Angiotensin II receptor blockers or thiazide-type diuretics other than study medication.
  * Over-the-counter products not permitted by investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 837 (Actual)
Dates: Start 2009-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Executive Medical Director, Clinical Science, Study Director — Takeda
Locations (26):
- Graz, Styria, Austria
- Germany (3):
  - Karlsruhe, Baden-Wurttemberg
  - Hanover, Lower Saxony
  - Kiel-Kronshagen, Schleswig-Holstein
- Netherlands (8):
  - Breda, North Brabant
  - Eindhoven, North Brabant
  - Amsterdam, North Holland
  - Groningen, Provincie Groningen
  - Velp, Rheden
  - Leiderdorp, South Holland
  - Rotterdam, South Holland
  - Zoetermeer, South Holland
- Poland (7):
  - Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Skierniewice, L0dz
  - Zgierz, L0dz
  - Gdansk, Pomeranian
  - Gdynia, Pomeranian
  - Sopot, Pomeranian
  - Mikołów, Silesian
- United Kingdom (7):
  - Avon, England
  - Bolton, England
  - Chorley, England
  - Inverness, England
  - Liverpool, England
  - Surrey, England
  - Warwickshire, England

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 79 investigative sites in the United States, Netherlands, Poland, the United Kingdom and Germany from 27 October 2009 to 17 November 2011.
Pre-assignment Details: Participants with a diagnosis of essential hypertension were randomized to receive open-label treatment with either Azilsartan Medoxomil and Chlorthalidone or Olmesartan Medoxomil and Hydrochlorothiazide for up to 52 weeks.
Groups:
- Azilsartan Medoxomil and Chlorthalidone: Azilsartan medoxomil 40 mg and chlorthalidone 12.5 mg combination tablet, orally, once daily for up to 52 weeks. For participants who did not achieve target blood pressure by Week 4, titration to a maximum dose of azilsartan medoxomil 80 mg and chlorthalidone 25 mg. Additional antihypertensive agents could be added as needed to achieve blood pressure control.
- Olmesartan Medoxomil and Hydrochlorothiazide: Participants in the United States: Olmesartan medoxomil 20 mg and hydrochlorothiazide 12.5 mg combination tablet, orally, once daily for up to 52 weeks. For participants who did not achieve target blood pressure by Week 4, titration to a maximum dose of Olmesartan medoxomil 40 mg and hydrochlorothiazide 25 mg. Participants in Europe: Olmesartan medoxomil 20 mg and hydrochlorothiazide 12.5 mg combination tablet, orally, once daily for up to 52 weeks. For participants who did not achieve target blood pressure by Week 4, titration to a maximum dose of Olmesartan medoxomil 20 mg and hydrochlorothiazide 25 mg. Additional antihypertensive agents could be added as needed to achieve blood pressure control.
Period: Overall Study
Arm/Group | Azilsartan Medoxomil and Chlorthalidone | Olmesartan Medoxomil and Hydrochlorothiazide
Started | 418 | 419
Completed | 287 | 330
Not Completed | 131 | 89
Not completed — Adverse Event | 75 | 37
Not completed — Major Protocol Deviation | 6 | 7
Not completed — Lost to Follow-up | 14 | 16
Not completed — Withdrawal by Subject | 31 | 20
Not completed — Lack of Efficacy | 0 | 2
Not completed — Other | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azilsartan Medoxomil and Chlorthalidone | Olmesartan Medoxomil and Hydrochlorothiazide | Total
Number analyzed (Participants) | 418 | 419 | 837
Age Continuous [Mean (Standard Deviation); unit: years] | 58.5 (10.79) | 57.6 (10.80) | 58.1 (10.80)
Age, Customized [Number; unit: participants]
  <45 years | 46 | 48 | 94
  45 to 64 years | 251 | 259 | 510
  65 to 74 years | 94 | 93 | 187
  ≥75 years | 27 | 19 | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 192 | 173 | 365
  Male | 226 | 246 | 472
Race/Ethnicity, Customized [Number; unit: participants] — Ethnicity was only collected from U.S. sites.
  participants
    Hispanic or Latino | 40 | 41 | 81
    Non-Hispanic or Latino | 209 | 205 | 414
    Not collected | 169 | 172 | 341
    Missing | 0 | 1 | 1
Race/Ethnicity, Customized [Number; unit: participants] — Participants could choose more than 1 category for race. Participants who choose more than 1 race category are included in each category indicated and are also included in the multiracial category.
  participants
    American Indian or Alaska Native | 4 | 5 | 9
    Asian | 4 | 7 | 11
    Black or African American | 72 | 74 | 146
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    White | 341 | 336 | 677
    Multiracial | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  Poland | 52 | 54 | 106
  United States | 249 | 247 | 496
  Netherlands | 56 | 58 | 114
  Germany | 22 | 21 | 43
  United Kingdom | 39 | 39 | 78
Height [Mean (Standard Deviation); unit: cm] | 169.9 (10.2) | 169.6 (10.1) | 169.8 (10.1)
Weight [Mean (Standard Deviation); unit: kg] | 91.00 (21.025) | 92.00 (21.727) | 91.50 (21.373)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.4 (6.21) | 31.9 (6.63) | 31.7 (6.42)
Smoking history [Number; unit: participants]
  Never smoked | 214 | 205 | 419
  Current smoker | 82 | 78 | 160
  Ex-smoker | 122 | 136 | 258
Diabetes Status [Number; unit: participants]
  Yes | 64 | 59 | 123
  No | 354 | 360 | 714
Estimated glomerular filtration rate [Number; unit: participants]
  Moderate impairment: ≥30 and <60 ml/min/1.73 m^2 | 54 | 43 | 97
  Mild impairment: ≥60 and <90 ml/min/1.73 m^2 | 275 | 265 | 540
  Normal: ≥90 ml/min/1.73 m^2 | 87 | 110 | 197
  Missing | 2 | 1 | 3
Chronic Kidney Disease (CKD) status [Number; unit: participants] — Participants were considered to have CKD if their estimated glomerular filtration rate (GFR) was <60 mL/min/1.73 m^2 or urinary albumin:creatinine ratio (UACR) was >200 mg albumin/g creatinine at Screening.
  participants
    Yes | 59 | 51 | 110
    No | 359 | 368 | 727
Systolic blood pressure [Number; unit: participants]
  ≥140 - < 160 mmHg | 1 | 1 | 2
  ≥160 - < 180 mmHg | 382 | 385 | 767
  ≥180 mm Hg | 35 | 33 | 68
Diastolic blood pressure [Number; unit: participants]
  < 90 mmHg | 107 | 103 | 210
  ≥90 mmHg | 311 | 316 | 627

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least 1 Adverse Event
Description: An adverse event is defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product without regard to causality.
Time Frame: From Week 0 (Day 1) to Week 52.
Population: Safety analysis set: All participants who received at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil and Chlorthalidone | Olmesartan Medoxomil and Hydrochlorothiazide
Number analyzed (Participants) | 418 | 419
percentage of participants | 78.5 | 76.4

2. Secondary Outcome: Percentage of Participants With Serum Creatinine Elevations Greater Than 50% From Baseline and Greater Than the Upper Limit of Normal (ULN)
Description: Serum creatinine was measured at every visit and evaluated as a laboratory parameter of special interest. The percentage of participants with creatinine increase ≥50% from Baseline and greater than ULN was summarized: - At any visit (includes transient and persistent elevations). - At the Final Visit (includes persistent elevations and participants whose first elevation may have been at the Final Visit). - At least 2 consecutive visits (includes only persistent elevations).
Time Frame: Baseline and Week 52
Population: Safety analysis set.
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil and Chlorthalidone | Olmesartan Medoxomil and Hydrochlorothiazide
Number analyzed (Participants) | 418 | 419
percentage of participants
  At any postbaseline visit | 14.2 | 5.8
  at the Final Visit | 5.9 | 1.0
  ≥2 consecutive elevations | 5.1 | 1.2

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 14 days (or 30 days for a serious adverse event) after the last dose of study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Azilsartan Medoxomil and Chlorthalidone | Olmesartan Medoxomil and Hydrochlorothiazide
Serious Adverse Events (participants affected / at risk) | 24/418 | 26/419
Other Adverse Events (participants affected / at risk) | 217/418 | 183/419
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan Medoxomil and Chlorthalidone (N=418) | Olmesartan Medoxomil and Hydrochlorothiazide (N=419)
Angina pectoris (Cardiac disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Hemorrhoid (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 2
Drowning (General disorders) | 1 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0
Cholelitiasis (Hepatobiliary disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2
Septic shock (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Rectal abscess (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 2
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Skeletal injury (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound secretion (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Syncope (Nervous system disorders) | 2 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Radicular syndrome (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Major depression (Psychiatric disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Rectocele (Reproductive system and breast disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan Medoxomil and Chlorthalidone (N=418) | Olmesartan Medoxomil and Hydrochlorothiazide (N=419)
Diarrhoea (Gastrointestinal disorders) | 20 | 21
Nausea (Gastrointestinal disorders) | 20 | 21
Fatigue (General disorders) | 21 | 17
Nasopharyngitis (Infections and infestations) | 51 | 48
Upper respiratory tract infection (Infections and infestations) | 20 | 27
Blood creatinine increased (Investigations) | 90 | 35
Dizziness (Nervous system disorders) | 68 | 53
Headache (Nervous system disorders) | 31 | 46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.